CLINICAL TRIAL: NCT00553254
Title: A PHASE 1/2, OPEN-LABEL, SINGLE ARM TRIAL TO DETERMINE THE RECOMMENDED PHASE 2 DOSE AND EVALUATE THE EFFICACY OF PF-00299804 IN PATIENTS IN KOREA WITH KRAS WILD TYPE ADVANCED NSCLC, WHICH IS REFRACTORY TO CHEMOTHERAPY AND ERLOTINIB OR GEFITINIB
Brief Title: Trial Of PF-00299804 In Patients With Advanced Refractory Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471003
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Carcinoma, Non Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: PF-00299804 — Single arm (no comparator) study, oral once daily dosing, dose escalation (it is a phase 1/2 study) until disease progression, unacceptable toxicity or withdrawal of consent

SUMMARY:
To assess the safety and efficacy of PF-00299804 in patients with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* Prior treatment with and failure of at least one regimen of chemotherapy and erlotinib or gefitinib
* Prior treatment with no more than two chemotherapy regimens, including adjuvant treatment
* Measurable disease

Exclusion Criteria:

* Chemotherapy, radiotherapy, biological or investigational agents within 4 weeks of baseline disease assessment
* Patients who lack of tolerance of erlotinib therapy
* Patients with known brain Metastases
* Patients with demonstrated history of or presence of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-02-05 (Actual); Primary Completion 2010-08-03 (Actual); Study Completion 2014-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- South Korea (3):
  - Seoul National University Hospital, Department of Internal Medicine, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Yonsei Cancer Center, Seoul
  - Samsung Medical Center, Department of Medicine, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Park K, Cho BC, Kim DW, Ahn MJ, Lee SY, Gernhardt D, Taylor I, Campbell AK, Zhang H, Giri N, Letrent SP, O'Connell J, Heo DS. Safety and efficacy of dacomitinib in korean patients with KRAS wild-type advanced non-small-cell lung cancer refractory to chemotherapy and erlotinib or gefitinib: a phase I/II trial. J Thorac Oncol. 2014 Oct;9(10):1523-31. doi: 10.1097/JTO.0000000000000275. PMID 25521398
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7471003&StudyName=Trial%20Of%20PF-00299804%20In%20Patients%20With%20Advanced%20Refractory%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-00299804 30 mg - Phase 1: A single dose of PF-00299804 30 milligram (mg) tablet orally on or before Day -9 followed by PF-00299804 30 mg tablet orally once daily continuously in 21-day cycles starting from Day 1 until unacceptable toxicity, disease progression, withdrawal from the trial, or death.
- PF-00299804 45 mg - Phase 1: A single dose of PF-00299804 45 mg tablet orally on or before Day -9 followed by PF-00299804 45 mg tablet orally once daily continuously in 21-day cycles starting from Day 1 until unacceptable toxicity, disease progression, withdrawal from the trial, or death.
- PF-00299804 45 mg - Phase 2: PF-00299804 45 mg tablet orally once daily continuously in 21-day cycles starting from Day 1 until unacceptable toxicity, disease progression, withdrawal from the trial, or death.
Period: Overall Study
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1 | PF-00299804 45 mg - Phase 2
Started | 6 | 6 | 43
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 43
Not completed — Death | 3 | 6 | 25
Not completed — Lost to Follow-up | 0 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2
Not completed — Study terminated by Sponsor | 0 | 0 | 1
Not completed — Other | 1 | 0 | 13

BASELINE CHARACTERISTICS:
Population: Data for baseline characteristics was pre-specified in statistical analysis plan to be analyzed and summarized per phase.
Groups:
- PF-00299804 - Phase 1 All Participants: A single dose of PF-00299804 30 mg or 45 mg tablet orally on or before Day -9 followed by PF-00299804 30 mg or 45 mg tablet orally once daily continuously in 21-day cycles starting from Day 1 until unacceptable toxicity, disease progression, withdrawal from the trial, or death.
- Total: Total of all reporting groups
Arm/Group | PF-00299804 - Phase 1 All Participants | PF-00299804 45 mg - Phase 2 | Total
Number analyzed (Participants) | 12 | 43 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.3) | 57.0 (8.7) | 56.0 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 23 | 32
  Male | 3 | 20 | 23

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) - Phase 1
Description: The highest dose at which less than (<) 33 percent (%) of participants experienced dose-limiting toxicities (DLT) was to be designated as the maximum tolerated dose (MTD) as well as the RP2D. DLT was defined as any of the following events: Grade 3/4 (severe or life-threatening/ disabling adverse event [AE]) nausea, vomiting, or diarrhea (despite the use of adequate/maximal medical intervention and/or prophylaxis); Grade greater than or equal to (>=) 3 (severe or life-threatening/disabling AE or death related to AE) non-hematological toxicity; delayed (which delayed scheduled treatment for >14 days) recovery from toxicity related to treatment with PF-00299804; Grade 4 neutropenia (absolute neutrophil count [ANC] <500 cells per cubic millimeter [cells/mm^3] for 5 or more consecutive days or febrile neutropenia [fever >=38.5 degrees Celsius with ANC <1000 cells/mm^3]); and Grade 4 thrombocytopenia (<25,000 cells/mm^3) or bleeding which required platelet transfusion.
Time Frame: Baseline up to Day 21
Population: As-treated population included all enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg
Arm/Group | PF-00299804 - Phase 1 All Participants
Number analyzed (Participants) | 12
mg | 45

2. Primary Outcome: Progression-Free Survival (PFS) at Month 4 (PFS4m) - Phase 2
Description: PFS4m was defined as percent chance of being event free (event defined as progressive disease [PD] or death due to any cause, whichever occurred first) at 4 months. Progression was defined using Response Evaluation Criteria in Solid Tumors (RECIST), as at least 20 percent (%) increase in the sum of longest dimensions (LD) of target lesions, taking as reference the smallest sum of LD recorded since the treatment started and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Month 4
Population: Full analysis set (FAS) included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percent chance of being event-free
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 43
percent chance of being event-free | 47.2 [31.6 to 61.3]

3. Secondary Outcome: Progression-Free Survival (PFS) at Month 6 (PFS6m) - Phase 2
Description: PFS6m was defined as percent chance of being event free (event defined as PD or death due to any cause, whichever occurred first) at 6 months. Progression was defined using RECIST, as at least 20% increase in the sum of longest dimensions (LD) of target lesions, taking as reference the smallest sum of LD recorded since the treatment started and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Month 6
Population: FAS included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percent chance of being event-free
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 43
percent chance of being event-free | 24.8 [12.9 to 38.7]

4. Secondary Outcome: Overall Survival (OS) at Month 6 (OS6m) - Phase 2
Description: OS6m was defined as percent chance of being alive at Month 6.
Time Frame: Month 6
Population: FAS included all enrolled participants.
Measure: Number (95% Confidence Interval); unit: percent chance of being alive
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 43
percent chance of being alive | 80.7 [65.1 to 89.9]

5. Secondary Outcome: Percentage of Participants With Objective Response - Phase 1
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of the longest dimensions (LDs) of target lesion, taking as reference the baseline sum LD, associated to non-progressive disease response for non-target lesions. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response.
Time Frame: Baseline until disease progression or initiation of new anti-cancer therapy or death, assessed every 2 (odd-numbered) cycles up to 12 months after end of treatment (EOT) (EOT: up to Day 506)
Population: Response-evaluable population included all enrolled participants who received at least 1 dose of study medication, had an adequate baseline tumor assessment, and had at least 1 on-study tumor assessment after first dosing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1
Number analyzed (Participants) | 6 | 6
percentage of participants | 0.0 [0.0 to 45.9] | 33.3 [4.3 to 77.7]

6. Secondary Outcome: Soluble Protein Biomarkers Level
Description: Blood specimens were analyzed at a sponsor-designated laboratory for analysis of shed proteins/receptors related to Human Epidermal Growth Factor Receptor (HER) signaling (epidermal growth factor receptor [EGFR], HER2). These measurements were determined by enzyme-linked immunosorbent assay (ELISA). The data for all Phase 1 participants was combined for this outcome.
Time Frame: Cycle 1 Day 1 (C1D1, Baseline), Day 1 of each odd-numbered cycle up to Cycle 17 for both Phase 1 and Phase 2
Population: Biomarker analysis set: all enrolled participants who had baseline samples submitted as per Institutional Review Board/Independent Ethics Committee approval and participant consent. Data was pre-specified in statistical analysis plan to be analyzed and summarized per phase. Number analyzed = participants evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-00299804 - Phase 1 All Participants | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 12 | 43
nanogram per milliliter (ng/mL)
  EGFR: C1D1 | 58.57 (7.498) | 57.41 (13.146)
  EGFR: C3D1: number analyzed (Participants) | 10 | 27
  EGFR: C3D1 | 47.46 (7.845) | 50.81 (11.465)
  EGFR: C5D1: number analyzed (Participants) | 3 | 21
  EGFR: C5D1 | 46.76 (5.395) | 58.87 (13.627)
  EGFR: C7D1: number analyzed (Participants) | 1 | 12
  EGFR: C7D1 | 48.58 (NA) — No measure of dispersion calculated as there is only 1 participant | 55.83 (19.34)
  EGFR: C9D1: number analyzed (Participants) | 1 | 9
  EGFR: C9D1 | 42.83 (NA) — No measure of dispersion calculated as there is only 1 participant | 50.32 (26.214)
  EGFR: C11D1: number analyzed (Participants) | 1 | 7
  EGFR: C11D1 | 40.98 (NA) — No measure of dispersion calculated as there is only 1 participant | 63.69 (28.908)
  EGFR: C13D1: number analyzed (Participants) | 1 | 5
  EGFR: C13D1 | 67.34 (NA) — No measure of dispersion calculated as there is only 1 participant | 73.26 (29.487)
  EGFR: C15D1: number analyzed (Participants) | 1 | 4
  EGFR: C15D1 | 52 (NA) — No measure of dispersion calculated as there is only 1 participant | 49.45 (14.358)
  EGFR: C17D1: number analyzed (Participants) | 1 | 4
  EGFR: C17D1 | 66.62 (NA) — No measure of dispersion calculated as there is only 1 participant | 57.95 (24.923)
  HER2: C1D1 | 9.51 (2.418) | 9.54 (5.859)
  HER2: C3D1: number analyzed (Participants) | 10 | 27
  HER2: C3D1 | 8.85 (1.125) | 8.36 (4.284)
  HER2: C5D1: number analyzed (Participants) | 3 | 21
  HER2: C5D1 | 9.63 (2.542) | 9.29 (5.138)
  HER2: C7D1: number analyzed (Participants) | 1 | 12
  HER2: C7D1 | 6.7 (NA) — No measure of dispersion calculated as there is only 1 participant | 11.57 (5.342)
  HER2: C9D1: number analyzed (Participants) | 1 | 9
  HER2: C9D1 | 5.6 (NA) — No measure of dispersion calculated as there is only 1 participant | 8.49 (4.124)
  HER2: C11D1: number analyzed (Participants) | 1 | 7
  HER2: C11D1 | 6.3 (NA) — No measure of dispersion calculated as there is only 1 participant | 8.2 (4.122)
  HER2: C13D1: number analyzed (Participants) | 1 | 5
  HER2: C13D1 | 11.7 (NA) — No measure of dispersion calculated as there is only 1 participant | 9.51 (5.97)
  HER2: C15D1: number analyzed (Participants) | 1 | 4
  HER2: C15D1 | 7.4 (NA) — No measure of dispersion calculated as there is only 1 participant | 5.43 (1.99)
  HER2: C17D1: number analyzed (Participants) | 1 | 4
  HER2: C17D1 | 8.9 (NA) — No measure of dispersion calculated as there is only 1 participant | 6.27 (2.626)

7. Secondary Outcome: Number of Participants With Epidermal Growth Factor Receptor (EGFR), Kirsten Rat Sarcoma (KRAS), and Human Epidermal Growth Factor Receptor-2 (HER2) Mutation Status
Description: Tumor tissue was analyzed at a sponsor-designated laboratory to investigate EGFR, KRAS and HER2 status (wild type or mutated). Participants who did not provide samples for central laboratory analysis confirmation were classified as "unknown". The data for all Phase 1 participants was combined for this outcome.
Time Frame: Screening
Population: Biomarker analysis set: all enrolled participants who had baseline samples submitted as per Institutional Review Board/Independent Ethics Committee approval and participant consent. Data was pre-specified in statistical analysis plan to be analyzed and summarized per phase.
Measure: Number; unit: participants
Arm/Group | PF-00299804 - Phase 1 All Participants | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 12 | 43
participants
  EGFR Status: Wild Type | 3 | 3
  EGFR Status: Mutant | 2 | 12
  EGFR Status: Unknown | 7 | 28
  KRAS Status: Wild Type | 9 | 29
  KRAS Status: Mutant | 0 | 0
  KRAS Status: Unknown | 3 | 14
  HER2 Status: Wild Type | 0 | 9
  HER2 Status: Mutant | 0 | 1
  HER2 Status: Unknown | 12 | 33

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-00299804 30 mg and PF-00299804 45 mg
Description: Data in "PF-00299804 45 mg" treatment arm at Cycle 0 Day -9 (C0D-9) represents participants from Phase 1 only and at C1D14 represents participants from both Phase 1 and Phase 2.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24, 72, 144, 216 hours post-dose on C0D-9 for Phase 1, 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C1D14 for Phase 1 and 2
Population: Pharmacokinetic (PK): all participants who received at least 1 dose of study drug and had at least 1 measured plasma concentration. "number analyzed"=participants evaluable for specified time-point. PK analysis was done by dose level instead of by phase. Participants started from the same dose level were combined together for PK analysis.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Groups:
- PF-00299804 45 mg: A single dose of PF-00299804 45 mg tablet orally on or before Day -9 followed by PF-00299804 45 mg tablet orally once daily continuously in 21-day cycles starting from Day 1 during Phase 1 or PF-00299804 45 mg tablet orally once daily continuously in 21-day cycles during Phase 2, until unacceptable toxicity, disease progression, withdrawal from the trial, or death.
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg
Number analyzed (Participants) | 6 | 40
nanogram per milliliter (ng/mL)
  C0D-9: number analyzed (Participants) | 6 | 6
  C0D-9 | 13.34 (4.8205) | 21.30 (12.356)
  C1D14 | 56.96 (20.572) | 82.71 (38.788)

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-00299804 30 mg and PF-00299804 45 mg
Description: Data in "PF-00299804 45 mg" treatment arm at C0D-9 represents participants from Phase 1 only and at C1D14 represents participants from both Phase 1 and Phase 2.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24, 72, 144, 216 hours post-dose on Cycle 0 Day -9 (C0D-9) for Phase 1, 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C1D14 for Phase 1 and 2
Population: PK analysis set included all participants who received at least 1 dose of study drug and had at least 1 measured plasma concentration. "number analyzed"=participants evaluable for specified time-point. PK analysis was done by dose level instead of by phase. Participants started from the same dose level were combined together for PK analysis.
Measure: Median (Full Range); unit: hours
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg
Number analyzed (Participants) | 6 | 40
hours
  C0D-9: number analyzed (Participants) | 6 | 6
  C0D-9 | 8.00 [4.17 to 24.0] | 4.96 [1.98 to 8.00]
  C1D14 | 5.03 [0.000 to 24.0] | 6.10 [0.000 to 24.0]

10. Secondary Outcome: Plasma Decay Half-Life (t1/2) of PF-00299804 30 mg and PF-00299804 45 mg - Phase 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24, 72, 144, 216 hours post-dose on Cycle 0 Day -9 (C0D-9)
Population: PK analysis set for Phase 1 included all participants who received at least 1 dose of study medication and had at least 1 measured plasma concentration.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1
Number analyzed (Participants) | 6 | 6
hours | 63.60 (30.271) | 54.02 (13.461)

11. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hour Post-Dose (AUC0-24) of PF-00299804 30 mg and PF-00299804 45 mg
Description: AUC0-24: Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours post dose. Data in "PF- 00299804 45 mg" treatment arm at C0D-9 represents participants from Phase 1 only and at C1D14 represents participants from both Phase 1 and Phase 2.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on Cycle 0 Day -9 (C0D-9) for Phase 1, 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C1D14 for Phase 1 and 2
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg
Number analyzed (Participants) | 6 | 40
nanogram*hour per milliliter (ng*hr/mL)
  C0D-9: number analyzed (Participants) | 6 | 6
  C0D-9 | 221.6 (87.063) | 354.8 (153.31)
  C1D14 | 1075 (515.66) | 1621 (664.87)

12. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-00299804 30 mg and PF-00299804 45 mg- Phase 1
Description: AUClast: Area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24, 72, 144, 216 hours post-dose on C0D-9
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 893.4 (516.50) | 1248 (522.11)

13. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-00299804 30 mg and PF-00299804 45 mg - Phase 1
Description: AUCinf: Area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24, 72, 144, 216 hours post-dose on C0D-9
Population: as for outcome 10
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1018 (593.51) | 1348 (599.34)

14. Secondary Outcome: Accumulation Ratio (Rac) of PF-00299804 30 mg and PF-00299804 45 mg - Phase 1
Description: Rac was calculated by dividing AUC0-24 (C1D14) by AUC0-24 (C0D-9).
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C0D-9, 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C1D14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1
Number analyzed (Participants) | 6 | 6
ratio | 5.265 (2.2958) | 5.682 (2.5752)

15. Secondary Outcome: Average Plasma Concentration (Cavg) of PF-00299804 30 mg and PF-00299804 45 mg
Description: Data in "PF-00299804 45 mg" treatment arm represents participants from both Phase 1 and Phase 2.
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C1D14 for Phase 1 and 2
Population: PK analysis set included all participants who received at least 1 dose of study drug and had at least 1 measured plasma concentration. PK analysis was done by dose level instead of by phase. Participants started from the same dose level were combined together for PK analysis.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg
Number analyzed (Participants) | 6 | 40
ng/mL | 44.78 (21.439) | 67.52 (27.643)

16. Secondary Outcome: Linearity Ratio (Rss) of PF-00299804 30 mg and PF-00299804 45 mg - Phase 1
Description: Rss was calculated by dividing AUC0-24 (C1D14) by AUCinf (C0D-9).
Time Frame: 0 (pre-dose), 2, 4, 6, 8, 24, 72, 144, 216 hours post-dose on C0D-9, 0 (pre-dose), 2, 4, 6, 8, 24 hours post-dose on C1D14
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1
Number analyzed (Participants) | 6 | 6
ratio | 1.093 (0.3100) | 1.442 (0.5661)

17. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Ctrough) of PF-00299804 30 mg and PF-00299804 45 mg
Description: Data in "PF-00299804 45 mg" treatment arm represents participants from both Phase 1 and Phase 2.
Time Frame: 0 hours (pre-dose) on C2D1, C3D1, C4D1
Population: PK analysis set included all participants who received at least 1 dose of study drug and had at least 1 measured plasma concentration. PK analysis was done by dose level instead of by phase. Participants started from the same dose level were combined together for PK analysis."number analyzed" = participants evaluable for specified time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg
Number analyzed (Participants) | 6 | 40
ng/mL
  C2D1: number analyzed (Participants) | 5 | 40
  C2D1 | 45.96 (31.061) | 65.11 (33.673)
  C3D1: number analyzed (Participants) | 6 | 31
  C3D1 | 46.52 (23.329) | 66.98 (32.354)
  C4D1: number analyzed (Participants) | 6 | 32
  C4D1 | 40.34 (24.527) | 69.75 (37.584)

18. Secondary Outcome: Number of Participants With Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) - Phase 2
Description: EORTC QLQ-C30: included global health status/quality of life (QoL), functional (Fn) scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Scores were averaged, transformed to 0-100 scale; higher score for Global Qol/Fn scales=better level of QoL/functioning or higher score for symptom scales/items=greater degree of symptoms. Overall scale change is categorized as Improved (if average scales change from baseline: for Global QoL/Fn scales >=10; for symptom scale/item <=-10), Worsened (if average scales change from baseline: for Global QoL/Fn scales <=-10; for symptom scale/item >=10), and Stable (if average scales change from baseline >-10 but <10 for Global QoL/Fn scales and symptom scale/item) and participants in each category are reported.
Time Frame: Baseline up to end of treatment (up to Day 889)
Population: FAS included all enrolled participants. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure.
Measure: Number; unit: participants
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 39
participants
  Global QoL: Improved | 5
  Global QoL: Worsened | 18
  Global QoL: Stable | 16
  Physical Functioning: Improved | 2
  Physical Functioning: Worsened | 20
  Physical Functioning: Stable | 17
  Role Functioning: Improved | 2
  Role Functioning: Worsened | 22
  Role Functioning: Stable | 15
  Cognitive Functioning: Improved | 4
  Cognitive Functioning: Worsened | 17
  Cognitive Functioning: Stable | 18
  Emotional Functioning: Improved | 2
  Emotional Functioning: Worsened | 16
  Emotional Functioning: Stable | 21
  Social Functioning: Improved | 6
  Social Functioning: Worsened | 15
  Social Functioning: Stable | 18
  Fatigue: Improved | 3
  Fatigue: Worsened | 20
  Fatigue: Stable | 16
  Pain: Improved | 8
  Pain: Worsened | 15
  Pain: Stable | 16
  Nausea and Vomiting: Improved | 4
  Nausea and Vomiting: Worsened | 10
  Nausea and Vomiting: Stable | 25
  Dyspnea: Improved | 7
  Dyspnea: Worsened | 16
  Dyspnea: Stable | 16
  Loss of Appetite: Improved | 6
  Loss of Appetite: Worsened | 24
  Loss of Appetite: Stable | 9
  Insomnia: Improved | 9
  Insomnia: Worsened | 12
  Insomnia: Stable | 18
  Constipation: Improved | 9
  Constipation: Worsened | 8
  Constipation: Stable | 22
  Diarrhea: Improved | 0
  Diarrhea: Worsened | 36
  Diarrhea: Stable | 3
  Financial Difficulties: Improved | 10
  Financial Difficulties: Worsened | 9
  Financial Difficulties: Stable | 20

19. Secondary Outcome: Number of Participants With Change in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13) - Phase 2
Description: EORTC QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Scores averaged, transformed to 0-100 scale; higher symptom score = greater degree of symptoms. Overall scale change is categorized as Improved (if average scales change from baseline <=-10), Worsened (if average scales change from baseline >=10), and Stable (if average scales change from baseline >-10 but <10) and participants in each category are reported.
Time Frame: Baseline up to end of treatment (up to Day 889)
Population: FAS included all enrolled participants. Here "N" (number of participants analyzed) signifies participants who were evaluable for this measure. Medicine for pain was not summarized because a more comprehensive and reliable summary of concomitant medications was reported separately.
Measure: Number; unit: participants
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 39
participants
  Dyspnoea: Improved | 10
  Dyspnoea: Worsened | 16
  Dyspnoea: Stable | 13
  Coughing: Improved | 9
  Coughing: Worsened | 11
  Coughing: Stable | 19
  Haemoptysis: Improved | 0
  Haemoptysis: Worsened | 5
  Haemoptysis: Stable | 34
  Sore mouth: Improved | 1
  Sore mouth: Worsened | 33
  Sore mouth: Stable | 5
  Dysphagia: Improved | 4
  Dysphagia: Worsened | 19
  Dysphagia: Stable | 16
  Peripheral: Improved | 9
  Peripheral: Worsened | 10
  Peripheral: Stable | 20
  Alopecia: Improved | 7
  Alopecia: Worsened | 11
  Alopecia: Stable | 21
  Pain in chest: Improved | 10
  Pain in chest: Worsened | 10
  Pain in chest: Stable | 19
  Pain in arm or Shoulder: Improved | 16
  Pain in arm or Shoulder: Worsened | 11
  Pain in arm or Shoulder: Stable | 12
  Pain in other parts: Improved | 10
  Pain in other parts: Worsened | 14
  Pain in other parts: Stable | 15

20. Secondary Outcome: Dermatology Life Quality Index (DLQI) Total Score - Phase 2
Description: DLQI: 10-item questionnaire to measure how much the participant's skin problem has impacted their life over the previous week. All questions were answered on a 4-point Likert scale ranging from 0 (not at all/not relevant) to 3 (very much/prevented work or studying). The DLQI was calculated by summing the score of each question and ranged from 0 to 30, where higher scores indicate more quality of life impairment.
Time Frame: C1D1 (baseline), D1 of each subsequent cycle up to C44
Population: FAS included all enrolled participants. Here "number analyzed" signifies participants who were evaluable for specified time-point for each treatment arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 43
units on a scale
  C1D1 | 0.81 (1.99)
  C2D1: number analyzed (Participants) | 39
  C2D1 | 6.54 (5.51)
  C3D1: number analyzed (Participants) | 35
  C3D1 | 9.51 (7.88)
  C4D1: number analyzed (Participants) | 27
  C4D1 | 10.85 (7.49)
  C5D1: number analyzed (Participants) | 25
  C5D1 | 11.04 (6.77)
  C6D1: number analyzed (Participants) | 21
  C6D1 | 10.76 (8.04)
  C7D1: number analyzed (Participants) | 19
  C7D1 | 9.47 (6.27)
  C8D1: number analyzed (Participants) | 13
  C8D1 | 9.92 (5.56)
  C9D1: number analyzed (Participants) | 12
  C9D1 | 9.58 (4.44)
  C10D1: number analyzed (Participants) | 9
  C10D1 | 10.22 (6.10)
  C11D1: number analyzed (Participants) | 8
  C11D1 | 11.25 (6.09)
  C12D1: number analyzed (Participants) | 7
  C12D1 | 9.00 (4.36)
  C13D1: number analyzed (Participants) | 7
  C13D1 | 8.71 (6.05)
  C14D1: number analyzed (Participants) | 5
  C14D1 | 9.80 (6.76)
  C15D1: number analyzed (Participants) | 5
  C15D1 | 9.60 (5.94)
  C16D1: number analyzed (Participants) | 4
  C16D1 | 9.25 (7.04)
  C17D1: number analyzed (Participants) | 4
  C17D1 | 11.50 (10.28)
  C18D1: number analyzed (Participants) | 4
  C18D1 | 9.00 (7.07)
  C19D1: number analyzed (Participants) | 4
  C19D1 | 8.75 (6.18)
  C20D1: number analyzed (Participants) | 4
  C20D1 | 7.00 (6.48)
  C21D1: number analyzed (Participants) | 4
  C21D1 | 7.00 (6.98)
  C22D1: number analyzed (Participants) | 4
  C22D1 | 7.75 (5.56)
  C23D1: number analyzed (Participants) | 4
  C23D1 | 7.75 (5.50)
  C24D1: number analyzed (Participants) | 2
  C24D1 | 10.00 (2.83)
  C25D1: number analyzed (Participants) | 2
  C25D1 | 11.00 (1.41)
  C26D1: number analyzed (Participants) | 1
  C26D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C27D1: number analyzed (Participants) | 1
  C27D1 | 13.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C28D1: number analyzed (Participants) | 1
  C28D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C29D1: number analyzed (Participants) | 1
  C29D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C30D1: number analyzed (Participants) | 1
  C30D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C31D1: number analyzed (Participants) | 1
  C31D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C32D1: number analyzed (Participants) | 1
  C32D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C33D1: number analyzed (Participants) | 1
  C33D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C34D1: number analyzed (Participants) | 1
  C34D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C35D1: number analyzed (Participants) | 1
  C35D1 | 14.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C36D1: number analyzed (Participants) | 1
  C36D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C37D1: number analyzed (Participants) | 1
  C37D1 | 10.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C38D1: number analyzed (Participants) | 1
  C38D1 | 11.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C39D1: number analyzed (Participants) | 1
  C39D1 | 13.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C40D1: number analyzed (Participants) | 1
  C40D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C41D1: number analyzed (Participants) | 1
  C41D1 | 13.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C42D1: number analyzed (Participants) | 1
  C42D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C43D1: number analyzed (Participants) | 1
  C43D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.
  C44D1: number analyzed (Participants) | 1
  C44D1 | 12.00 (NA) — No measure of dispersion calculated as there is only 1 participant.

21. Secondary Outcome: Best Overall Response (BOR) - Phase 2
Description: Number of participants with BOR according to RECIST: CR= disappearance of all target and non-target lesions. PR= at least 30% decrease in sum of LDs of target lesion, taking as reference baseline sum LD, associated to non-progressive disease response for non-target lesions. Stable/no response= neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Objective progression= at least a 20% increase in sum of LDs of target lesions, taking as reference the smallest sum of LD recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Baseline until disease progression or initiation of new anti-cancer therapy or death, assessed every 2 (odd-numbered) cycles up to 12 months after EOT (EOT: up to Day 1723)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 41
participants
  Complete Response | 0
  Partial Response | 7
  Stable/No Response | 21
  Objective Progression | 13
  Indeterminate | 0

22. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from first documentation of objective tumor response to objective tumor progression or death due to any cause, whichever occurred first. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to any cause minus the date of the first CR or PR [which ever occurred first] that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: Baseline until disease progression or initiation of new anti-cancer therapy or death, assessed every 2 (odd-numbered) cycles up to 12 months after EOT (EOT: up to Day 506 for Phase 1 and up to Day 1723 for Phase 2)
Population: Analysis population included sub-set of participants from response-evaluable population, who had a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1 | PF-00299804 45 mg - Phase 2
Number analyzed (Participants) | 0 | 2 | 7
weeks |  | 41.9 [15.1 to 68.7] | 60.6 [10.1 to NA] — The upper limit of 95% confidence interval was not reached.

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time that the participant provided informed consent through and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-00299804 30 mg - Phase 1 | PF-00299804 45 mg - Phase 1 | PF-00299804 45 mg - Phase 2
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 9/43
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 30 mg - Phase 1 (N=6) | PF-00299804 45 mg - Phase 1 (N=6) | PF-00299804 45 mg - Phase 2 (N=43)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 5
Pneumonia (Infections and infestations) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-00299804 30 mg - Phase 1 (N=6) | PF-00299804 45 mg - Phase 1 (N=6) | PF-00299804 45 mg - Phase 2 (N=43)
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 4
Constipation (Gastrointestinal disorders) | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 6 | 36
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 6
Nausea (Gastrointestinal disorders) | 1 | 2 | 7
Stomatitis (Gastrointestinal disorders) | 2 | 3 | 20
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Asthenia (General disorders) | 0 | 0 | 3
Chest discomfort (General disorders) | 0 | 1 | 2
Chest pain (General disorders) | 1 | 1 | 3
Fatigue (General disorders) | 0 | 0 | 8
Mucosal inflammation (General disorders) | 2 | 3 | 7
Pyrexia (General disorders) | 0 | 0 | 3
Xerosis (General disorders) | 0 | 1 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 2
Paronychia (Infections and infestations) | 3 | 3 | 29
Pneumonia (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3
Headache (Nervous system disorders) | 1 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 6 | 35
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 16
Hair disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 3 | 13
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 15
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 5
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.